CLINICAL TRIAL: NCT04402905
Title: Observational Study in Diagnosed Patients Covid-19, Supported on an Outpatient Basis.
Brief Title: Observational Study in Diagnosed Patients COVID-19, Supported on an Outpatient Basis. (COVID-PSL)
Acronym: COVID-PSL
Status: Completed | Type: Observational
Sponsor: Centre de Recherches et d'Etude sur la Pathologie Tropicale et le Sida (Other)
Responsible Party: Sponsor
Other Study IDs: CREPATS 011
Record Dates: First submitted 2020-05-20; First posted 2020-05-27 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Coronavirus Infection
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COVID-19 is an infection linked to a new coronavirus: SARS-CoV-2, which appeared in Wuhan in China at the end of 2019, and which has since spread around the world, responsible for a new major pandemic, which is upsetting the whole world.

If severe respiratory disease is the form that constitutes the extreme gravity of the disease (mortality, with more than 170,000 deaths worldwide to date).

However, there is a great heterogeneity of clinical forms with asymptomatic or symptomatic pauci forms, moderate forms, up to severe forms.

Different symptoms may appear: fever, cough, asthenia, dyspnea, gastrointestinal forms, anosmia and / or ageusia, skin involvement, etc.

Given the novelty of this infection, several questions remain:

* What are all the symptoms that can be contracted by a COVID-19 patient?
* Are there clinical forms not described?
* What is the evolutionary profile, the healing time of this disease in patients treated on an outpatient basis?
* What are the factors associated with a prolonged form of COVID-19 disease, including on an outpatient basis?

DETAILED DESCRIPTION:
Most of the descriptive studies relating to COVID-19 relate to the severe forms of the disease managed in the hospital sector.

Few data have been published on moderate forms, requiring no hospitalization, of strict outpatient management.

These so-called moderate forms, however, constitute the majority of cases of COVID-19 (approximately 80%).

In the Infectious and Tropical Diseases Department of Pitie Salpetriere, COVIDOM pilot site, at the beginning of March, during the intensification of the epidemic in France, a weekly telephone consultation was set up to take care of people tested for COVID + by PCR, or people not tested by PCR, or even tested with negative PCR but symptomatic and followed at home, suffering from moderate form of COVID-19, as well as their contact cases if they wished.

Telemedicine is particularly suitable in this epidemic context, ensuring continuity of care, while limiting face-to-face consultations, thus reducing the risk of cross-contamination.

Given the novelty of this infection, it is important to be able to best characterize these ambulatory forms, as well as their evolution, in order to manage these patients, and to offer primary care physicians a more detailed description of these forms. , which they are and will be called upon to take care of, general medicine being central to dealing with the epidemic.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* COVID PCR + patient: Patient screened positive by PCR on nasopharyngeal swab
* or COVID-like patient: Patient not screened, but considered COVID + because contact with a COVID PCR + person, and presenting symptoms suggestive of COVID-19 among:
* Influenza-like illness (fever, body aches, arthralgia, etc.)
* Respiratory form: dyspnea, cough, rhinitis
* Gastrointestinal form: diarrhea, nausea, vomiting
* Anosmia and / or ageusia
* or patient COVID PCR-: If patient tested negative by PCR on nasopharyngeal swab, but showing signs suggestive of COVID-19.

Exclusion Criteria:

* Patient objecting to the use of their data for research purposes
* Patient under justice or deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrolment will be done from the active queue of patients included in the COVIDOM / PSL platform.
  This study will be a monocentric data collection. The patient is called, on working days, weekly from D0 to D30, and beyond if the symptoms persist on D30.
  Data will be collected at D0, D7, D14, D21 and D30. The visit on D30 corresponds to the end of the systematic weekly telephone interviews if the patient has reached complete recovery, defined by the absence of symptoms for 3 days.
  If the symptoms persist on D30: monitoring is continued, on D45 and D60, and beyond if necessary.
Sampling Method: Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
COVID-PSL Cohort | 3 months
  measure of the absence of symptoms to assess the rate of complete clinical recovery on day 30

CONTACTS AND LOCATIONS:
Overall Officials: Christine Katlama, MD, Principal Investigator — Pitie-Salpetriere Hospital
Locations (1):
- Yasmine Dudoit, Paris, France